CLINICAL TRIAL: NCT06645925
Title: Novel Soft Tissue Augmentation Technique Using Free Gingival Graft Simultaneous With Implant Placement in Posterior Mandible: A 1-year Randomized Clinical Trial
Brief Title: Novel Soft Tissue Augmentation Technique Using Free Gingival Graft Simultaneous With Posterior Mandibular Implant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Collaborators: International Dental Contiuing Education (Network)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, CEO and Clinical Director, International Dental Contiuing Education
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDCE - 13
Record Dates: First submitted 2024-09-05; First posted 2024-10-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Free Gingival Graft; Free Gingival Graft Volume Change; Keratinized Tissue
Keywords: FGG; Delayed implant placement; Keratinized mucosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One Step Protocol (Experimental): FGG simultaneous with delayed implant placement
  Interventions: Procedure: One Step Protocol
- Two Steps protocol (Active Comparator): Conventional FGG protocol, prior to implant placement
  Interventions: Procedure: Two Steps Protocol

INTERVENTIONS:
Procedure: One Step Protocol — FGG will be done simultaneous with implant placement
  Arms: One Step Protocol
Procedure: Two Steps Protocol — Conventional FGG protocol, prior to implant placement
  Arms: Two Steps protocol

SUMMARY:
Presence of keratinized tissue (KT) around dental implants, plays a crucial role in stability and health of peri-implant tissues. Several studies reported that, minimum of 2 mm keratinized tissue width is required to achieve long-term longevity. Insufficient keratinized mucosa leads to biofilm accumulation, soft tissue inflammation, eventually peri-implant mucositis and peri-implantitis. Hence, the aim of the present trial is to evaluate KTW gain, linear and volumetric changes in buccal soft tissue along with hard tissue alterations following implant restoration at sites treated either with delayed implant placement & simultaneous FGG or the conventional FGG protocol prior to implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Adults at or above the age of 18.
* Lower Posterior missing tooth/ teeth with minimal KT < 2mm
* Sufficient alveolar ridge length minimum 13-15 mm to IAN

  •. Sufficient alveolar ridge width minimum of 6 mm
* Patients able to tolerate surgical periodontal procedures.
* Patients who provided an informed consent and accepted the one-year follow-up period.

Exclusion Criteria

* Patients diagnosed with periodontal diseases (Caton et al., 2018).
* Current or previous smokers.
* Pregnant and lactating females.
* Patients with medical conditions that would compromise the surgical procedures; uncontrolled diabetes mellitus, taking intravenous Bisphosphonates for treatment of osteoporosis.
* Patients with active infection related to the site of implant.
* Patients with parafunctional habits.
* Patients with shallow vestibule

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Keratinized tissue width | 0 - 3 - 6 - 12 months
  Measure Clinically and Digitally at 0 - 3 - 6 - 12 months postoperative

SECONDARY OUTCOMES:
Linear changes in buccal soft tissue contour | 0-3, 0-6, 0-12 Months
Interdental Papilla height changes | 12 months
Midfacial margin changes | 12 Months
Crestal bone level changes | 12 Months
Bone labial to the implant | 12 Months
Survival Rate | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Continuing Education, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No